CLINICAL TRIAL: NCT05139160
Title: Aminoacidemia and Protein Kinetics in Response to the Ingestion of Plant-based Protein Blends
Acronym: PBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14040
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Nutrition, Healthy
Keywords: plant-based protein; whey protein; protein quality; muscle protein synthesis

STUDY DESIGN:
Intervention Model Description: The study design will be a randomized, double blind, crossover trial.
Who Masked: Participant, Investigator
Masking Description: The study design will be a randomized, double blind, crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein isolate (Experimental): Whey protein isolate is the 'gold standard' of protein supplements due to being rich in essential amino acids and leucine. Leucine is a key amino acid the is required to stimulate muscle protein synthesis. Muscle protein synthesis is the major mechanism the underpins muscle growth. The whey protein would ostensibly serve as a positive control.
  Interventions: Dietary Supplement: Protein quality
- Plant based protein isolate (Experimental): Current plant-based protein isolates available contain insufficient amounts of leucine, and are less digestible, resulting in a reduced muscle protein synthesis responses. The plant based protein would ostensibly serve as a negative control.
  Interventions: Dietary Supplement: Protein quality
- Plant based protein isolate + leucine (Experimental): Enriching plant-based protein with leucine will increase the 'quality' of said protein source and theoretically should have similar muscle protein synthetic responses to whey protein.
  Interventions: Dietary Supplement: Protein quality

INTERVENTIONS:
Dietary Supplement: Protein quality — the present investigation aims to study a novel protein based protein isolate blend with and without leucine an compared with whey protein isolate to determine its impact aminoacidemia and muscle protein synthesis healthy adults.

SUMMARY:
The present investigation aims to study a novel plant based protein isolate blend to determine if it results in similar muscle building responses compared to whey protein isolate.

DETAILED DESCRIPTION:
Whey protein is considered the 'gold standard' to maintain body proteins (muscle, skin, bone). When isolated from milk, whey protein isolate (WPI) contains all nine essential amino acids (EAA) which are 'building blocks' that are needed to support the maintenance of body proteins. To date, there is no plant-based protein (PBP) isolate that compares to the recommended WPI towards how our body builds or supports our muscles. WPI is considered the 'gold standard' because it contains all of the EAA which provide the right amount of 'building blocks' to support our muscles. Current PBP isolates available contain insufficient amounts of EAA, and are less digestible, resulting in less 'building blocks' available to support our muscles. Recently, plant protein combinations have been designed to provide the right amounts of all the EAAs. Therefore, the aim of the present study is to determine the effects of a novel PBP blend on muscle protein synthesis responses by comparing it to WPI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between the ages of 18 - 30 years (inclusive)
2. Have a body mass index (BMI) between 18-30 kg·m2 (inclusive)
3. Be in general good health as assessed by a general health questionnaire
4. Non-smoking
5. Regular menstrual cycle and not using hormonal contraceptives
6. Willing and able to provide informed consent

Exclusion Criteria:

1. Currently using analgesic or anti-inflammatory drugs
2. A history of neuromuscular problems or muscle and/or bone wasting diseases
3. Any acute or chronic illness, metabolic disorders
4. Currently using corticosteroids
5. Use of hormonal contraceptives or anabolic steroids (e.g. testosterone)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis | Over a 5 hour period
  A marker of muscle growth

SECONDARY OUTCOMES:
Aminoacidemia | Over a 5 hour period
  Amino acids in the blood
Appetite and desire for specific food types in response to test drinks types H | Immediately before, and 30, 60, 120, 180 and 300 minutes after test drinks are consumed.
  Questionnaire on appetite and palpability of the drinks assessed by a visual analogue scale. 100 mm in length with words anchored at each end, expressing the most positive and the most negative rating used to assess hunger, satiety and fullness. Higher scores mean a better outcome.
Palatability of test drinks | Immediately after test drink are consumed.
  Questionnaire of palatability of test drinks assessed by a visual analogue scale. 100 mm in length with words anchored at each end, expressing the most positive and the most negative rating used to assess visual appeal, smell, taste, aftertaste and palatability. Higher scores mean a better outcome.
Questionnaire on safety | Over a 5 hour period
  Safety will be measured via a questionnaire; e.g. can the participant drink the test drinks and are they okay? Yes or no.
Tolerability of test drinks | Over a 5 hour period
  Tolerability will be measured using Visual Analog Scales anchored by the following descriptors: 0 - no symptoms at all; 100 - worst symptoms participant has ever experienced for the following: nausea, belching, feeling of fullness, vomiting, abdominal distension, flatulence, diarrhoea, dry mouth, and thirst.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Changhyun Lim, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim C, Janssen TAH, Currier BS, Paramanantharajah N, McKendry J, Abou Sawan S, Phillips SM. Muscle Protein Synthesis in Response to Plant-Based Protein Isolates With and Without Added Leucine Versus Whey Protein in Young Men and Women. Curr Dev Nutr. 2024 May 10;8(6):103769. doi: 10.1016/j.cdnut.2024.103769. eCollection 2024 Jun. PMID 38846451